CLINICAL TRIAL: NCT05006989
Title: Blueberry Intake and Infant Gut Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: U.S. Highbush Blueberry Council (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 20-1659
Record Dates: First submitted 2021-07-19; First posted 2021-08-16 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Infant Development
Keywords: Blueberries; Gut microbiota; Inflammation; Innate immunity; Early complementary feeding
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants will be provided pre-made whole blueberry freeze-dried powder to be consumed.
  Interventions: Other: Blueberry Powder
- Placebo Group (Placebo Comparator): Placebo powder with matching color and texture.
  Interventions: Other: Placebo Powder

INTERVENTIONS:
Other: Blueberry Powder — Administered one packet per day (10 grams/packet) and participants consume up to 10 grams per day.
  Arms: Intervention Group
Other: Placebo Powder — Administered one packet per day (10 grams/packet) and participants consume up to 10 grams per day.
  Arms: Placebo Group

SUMMARY:
The objective of this project is to investigate the effects of blueberries on gut microbiota, inflammation and innate immunity in breastfed infants during early complementary feeding (~5 to 12 months of age).

DETAILED DESCRIPTION:
Some details are intentionally left to out to preserve the scientific integrity of the study, and they will be included in the record after the study is completed.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy
* Full term (gestational age ≥ 37 weeks)
* No prior exposure of solid foods
* Exclusively breastfed (< 2 weeks of cumulative formula exposure)
* Willing to consume blueberry/placebo powder

Exclusion Criteria:

* Having health conditions that would affect normal growth
* Pre-term
* Consumed formula for more than two weeks
* Not willing to consume the blueberry/placebo powders

Ages: 4 Months to 5 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Gut Microbiome Composition Analyzed using 16S rRNA Amplicon Sequencing | Over 7 months
  16S rRNA amplicon sequencing is used to profile taxonomic makeup of fecal specimens. Within the gut microbiome composition, microbial diversity will be summarized using common ecological measures (Good's coverage, Sobs, and Shannon alpha diversity).
Infant Growth (Length) | Over 7 months
  Measured in cm
Infant Growth (Weight) | Over 7 months
  Measured in kg
Dietary Intake | Over 7 months
  3 day dietary recall with results generated by NDSR software

SECONDARY OUTCOMES:
Blueberry-Specific Food Signatures (Compounds) as Assessed by Metabolomics Analysis | Over 7 months
  Metabolomics analysis (nutri-metabolomics) is used to identify and validate food-derived biomarkers that may be classified as biomarkers of intake and/or biomarkers of effect, both of which can be linked to health indicators.

CONTACTS AND LOCATIONS:
Overall Officials: Minghua Tang, PhD, Principal Investigator — University of Colorado Denver | Anschutz
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Glime GNE, Matzeller KL, Frank DN, Kotter C, Kofonow JM, Robertson CE, Venter C, Campbell WW, Krebs NF, Tang M. Introducing blueberry powder as one of the first complementary foods changes the gut microbiota composition and diversity in U.S. human milk-fed infants: a double-blind, randomized controlled trial. Front Nutr. 2025 Sep 4;12:1623521. doi: 10.3389/fnut.2025.1623521. eCollection 2025. PMID 40977976